CLINICAL TRIAL: NCT01187563
Title: A Phase 4, Open-label, Repeat-Dose Study of the Safety and Pharmacodynamic Profile of Tocilizumab and Concomitant Methotrexate in Patients With Rheumatoid Arthritis
Brief Title: A Study of Tocilizumab in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-RA-1008
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis, tocilizumab
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an open-label, uncontrolled, observational study in patients with rheumatoid arthritis (RA) who are receiving tocilizumab concomitantly with methotrexate as part of their standard of care.

DETAILED DESCRIPTION:
This single arm, open label study evaluates the safety and pharmacodynamic profile of tocilizumab in RA patients. Participating patients are among those for whom tocilizumab is indicated and who are scheduled to receive tocilizumab as part of their normal care, in full compliance with the FDA-approved prescribing information. Study assessments consist of clinical evaluations and laboratory tests conducted in conjunction with the first three monthly intravenous infusions of tocilizumab. These assessments are designed to provide a better understanding of the pharmacodynamic effects and mechanistic actions of tocilizumab and help guide the clinical development of other therapeutic agents for RA. A total of 15 patients are expected to participate for approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Moderately to severely active rheumatoid arthritis
* Inadequate response to previous treatment with an anti-TNF agent
* Receiving methotrexate for at least 12 wks before study

Exclusion Criteria:

* Previous treatment with tocilizumab
* Previous treatment with other IL-6 receptor inhibitors
* Treatment with corticosteroids (oral prednisone >10 mg/day or equivalent) within 4 wks
* Conditions noted in the tocilizumab prescribing information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult rheumatoid arthritis patients with indication for treatment with tocilizumab.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety (clinical and laboratory parameters) | Throughout the study until week 10
  Proportion of patients with neutropenia, elevated transaminase, and/or decreased platelet count

SECONDARY OUTCOMES:
Treatment emergent adverse events | Throughout the study until week 10
  Post-baseline changes in vital signs, and hematological and biochemical parameters

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Worcester, Massachusetts
  - Duncansville, Pennsylvania